CLINICAL TRIAL: NCT06302699
Title: Clinical Utility of Ultrasensitive Chromosomal Aberrations Detection (UCAD) for Detecting Minimal Residual Disease (MRD) and Monitoring Clonal Evolution by Low-Pass Whole Genome Sequencing in Multiple Myeloma
Brief Title: Detecting Minimal Residual Diseases (MRD) and Monitoring Clonal Evolution Using Ultrasensitive Chromosomal Aberrations Detection (UCAD) in Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Suzhou Hongyuan Biotech Inc., Biobay, Suzhou, China. (Unknown)
Responsible Party: Principal Investigator, Gang An, Professor, Institute of Hematology & Blood Diseases Hospital, China
Other Study IDs: UCAD-MM-001
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: Minimal Residual Disease; Low-Pass Whole Genome Sequencing; Clonal Evolution; Ultrasensitive Chromosomal Aberrations Detection
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bone marrow mononuclear cells from multiple myeloma patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The presence of minimal residual disease (MRD) is an important prognostic factor for multiple myeloma, while copy number variation (CNV) is a widely accepted biomarker used for multiple myeloma (MM). Detecting MRD and monitoring clonal evolution by monitoring CNV using low-pass whole genome sequencing is promising due to its high analytical sensitivity. To evaluate the correlation between MRD detected by flow cytometry and low-pass whole genome sequencing, nearly 200 samples were collected for this study. We applied ultrasensitive chromosomal aberrations detection to detect CNV for each patient. The follow-up samples were then collected and sequencing used the same method.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with MM.
* With available baseline and sequential next-generation flow-MRD data.

Exclusion Criteria:

* Subjects without baseline and sequential next-generation flow-MRD data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple myeloma patients with baseline and sequential next-generation flow-MRD data are included in this study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Detection of copy number variation | From May 1, 2023 to December 31, 2023

SECONDARY OUTCOMES:
Serial monitoring of treatment response | From January 1, 2024 to May 31, 20224

CONTACTS AND LOCATIONS:
Locations (1):
- InsituteHBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng S, Ying Y, Xing N, Wang B, Qian Z, Zhou Z, Zhang Z, Xu W, Wang H, Dai L, Gao L, Zhou T, Ji J, Xu C. Noninvasive Detection of Urothelial Carcinoma by Cost-effective Low-coverage Whole-genome Sequencing from Urine-Exfoliated Cell DNA. Clin Cancer Res. 2020 Nov 1;26(21):5646-5654. doi: 10.1158/1078-0432.CCR-20-0401. Epub 2020 Oct 9. PMID 33037018